CLINICAL TRIAL: NCT02583009
Title: Multicenter, Randomized, Double-blind, Placebo-controlled Parallel-group, Dose Finding Phase II Clinical Trial to Evaluate Anti Rosacea Effect and Safety of PAC-14028 Cream (0.1%, 0.3%, 1.0%) in Rosacea Patients
Brief Title: A Study to Evaluate the Safety and Efficacy of PAC-14028 Cream in Rosacea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amorepacific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP-TRPV1_PII-03
Record Dates: First submitted 2015-09-30; First posted 2015-10-21 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PAC-14028 cream 0.1% (Experimental): PAC-14028 cream 0.1%, Twice daily for 4 weeks
  Interventions: Drug: PAC-14028 cream 0.1%
- PAC-14028 cream 0.3% (Experimental): PAC-14028 cream 0.3%, Twice daily for 4 weeks
  Interventions: Drug: PAC-14028 cream 0.3%
- PAC-14028 cream 1.0% (Experimental): PAC-14028 cream 1.0%, Twice daily for 4 weeks
  Interventions: Drug: PAC-14028 cream 1.0%
- PAC-14028 cream vehicle (Placebo Comparator): PAC-14028 cream vehicle, Twice daily for 4 weeks
  Interventions: Drug: PAC-14028 cream vehicle

INTERVENTIONS:
Drug: PAC-14028 cream 0.1% — Topical application
  Arms: PAC-14028 cream 0.1%
Drug: PAC-14028 cream 0.3% — Topical application
  Arms: PAC-14028 cream 0.3%
Drug: PAC-14028 cream 1.0% — Topical application
  Arms: PAC-14028 cream 1.0%
Drug: PAC-14028 cream vehicle — Topical application
  Arms: PAC-14028 cream vehicle

SUMMARY:
This clinical study is to determine the optimum dose of PAC-14028 cream in a therapeutic confirmatory clinical study by evaluating the safety and therapeutic equivalence of PAC-14028 cream 0.1%, 0.3% and 1.0% in patients with rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 19 - 70 years old
* Among the patients diagnosed with erythematotelangiectatic and papulopustular rosacea in accordance with the diagnostic criteria of the National Rosacea Society Expert Committee
* Subjects with rosacea scored 2 or more according to the Investigator Global Assessment (IGA) at screening

Exclusion Criteria:

* Those who can't be diagnosed or assessed for rosacea due to the presence of trauma, tattoo, scar, excessive hairs on the facial region
* Those who have received a facial laser treatment within 6 weeks
* Those who have been administered with oral retinoid or therapeutic vitamin A within 6 months
* Those who have received a hormonal treatment such as estrogen within 3 months
* Those who have been administered with systemic antibiotics or systemic steroid formulation within 4 weeks
* Those who have been administered with local retinoid, local steroid and local antibiotics and local medication for the treatment of rosacea on face within 4 weeks
* Those who have a history of blood disorder that can have a serious effect on the clinical study
* Women who are pregnant, lactating or who plan to be pregnant during the clinical study period or women of childbearing potential who do not use available contraceptive methods

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2014-10; Primary Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in Investigator Global Assessment (IGA) | Week 4 from the baseline
  Any intragroup and intergroup differences with respect to the IGA difference value on 28th day from the baseline.

SECONDARY OUTCOMES:
Improvement rate in Investigator Global Assessment (IGA) | Week 4 from the baseline
Change in the erythema severity score | Week 4 from the baseline
Rate of change in inflammatory lesion counts | Week 4 from the baseline
Change in erythema index | Week 4 from the baseline
Change in the telangiectasia severity score | Week 4 from the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Miyoung Park, PhD, Study Director — Amorepacific R&D Center
Locations (1):
- Korea University Ansan Hospital, Ansan-si, Gyeonggi-do, South Korea